CLINICAL TRIAL: NCT05382858
Title: Deep Brain Stimulation of the Posterior Subthalamic Area (PSA) Versus Subthalamic Nucleus (STN) for Tremor-dominant Parkinson's Disease: a Prospective, Randomized, Double-blinded, Cross-over Trial
Brief Title: PSA Versus STN DBS for TD-PD
Acronym: PSA-STN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Suzhou Sceneray Medical Co. , Ltd (Industry)
Responsible Party: Principal Investigator, LI DIANYOU, Doctor, Ruijin Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TDPSA
Record Dates: First submitted 2022-05-01; First posted 2022-05-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: tremor-dominant Parkinson's disease; deep brain stimulation; posterior subthalamic area; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSA-STN (Experimental): Participants randomized in this arm will receive bilateral PSA stimulation in the first two months in the randomized phase and then will be crossovered to the bilateral STN stimulation for another two months.
  Interventions: Device: Deep brain stimulation
- STN-PSA (Experimental): Participants randomized in this arm will receive bilateral STN stimulation in the first two months in the randomized phase and then will be crossovered to the bilateral PSA stimulation for another two months.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — active DBS with optimal stimulating parameters

SUMMARY:
The aim of this study is to compare the effectiveness of the deep brain stimulation in the posterior subthalamic area (PSA) versus the subthalamic nucleus (STN) for the treatment of tremor-dominant Parkinson's disease (PD) in a randomized, double-blinded, cross-over manner.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, crossover trial aiming at comparing the efficacy of PSA and STN DBS in treating tremor-dominant PD. Enrolled patients will undergo bilateral DBS surgery, targeting both PSA and STN with single trajectory. Two months post-implantation, patients enter a 4-month double-blinded crossover phase with PSA and STN DBS in randomized order. After 6 months post-implantation (at the end of the crossover phase), patients enter an open-label phase during which programming parameters are not restricted until the termination of the study at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease
* tremor-dominant subtype in the on-medication condition
* modified Hoehn-Yahr scale of 2 to 4 in the on-medication condition
* receiving regular anti-parkinsonian drugs for more than 6 weeks
* good compliance and written informed consent provided

Exclusion Criteria:

* Atypical parkinsonism
* History of stroke, encephalitis, neuroleptic uses, MRI scan with evidence of significant brain atrophy, lacunar infracts, or other conditions that might interfere with the intracranial surgery
* Presence of cognitive, or psychiatric or other co-morbidities (e.g., dementia, epilepsy, cranial traumatism, brain tumor, schizophrenia, severe depression or bipolar disorder, personality disorder, etc.) that might interfere with the patient's ability to complete the evaluations or to provide informed consent
* Presence of anatomical abnormalities in the target region
* Clinically significant medical history that would increase pre-/post-operative complications
* Other conditions considered by the investigators that might interfere with the surgery procedure, the follow-ups, and the interpretation of the data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the tremor sub-score of the Movement Disorder Society-sponsord Unified Parkinson's Disease Rating Scale Part III in the randomized phase | up to 6 months
  in the off-medication condition

SECONDARY OUTCOMES:
Change from baseline MDS UPDRS-III to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline MDS UPDRS-III to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline Fahn-Tolosa-Marin Clinical Rating Scale to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline Fahn-Tolosa-Marin Clinical Rating Scale to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline Timed up and go test (TUG) to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline Timed up and go test (TUG) to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline Berg balance scale to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline Berg balance scale to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
  in the off-medication condition
Change from baseline 39-item Parkinsons disease questionnaire to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline 39-item Parkinsons disease questionnaire to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline Levodopa equivalent daily dose to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline Levodopa equivalent daily dose to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline maximal phonatory time to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline maximal phonatory time to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline dysphonia severity index to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline dysphonia severity index to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline Mini-Mental Status Exam to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline Mini-Mental Status Exam to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline Beck depression inventory to the end of PSA stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Change from baseline Beck depression inventory to the end of STN stimulation phase in the randomization phase | up to 6 months (4-6 months depending on randomization arm)
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the MDS UPDRS-III in the randomized phase | up to 6 months
  in the off-medication condition
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the Fahn-Tolosa-Marin Clinical Rating Scale in the randomized phase | up to 6 months
  in the off-medication condition
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the Timed up and go test (TUG) in the randomized phase | up to 6 months
  in the off-medication condition
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the Berg balance scale in the randomized phase | up to 6 months
  in the off-medication condition
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the 39-item Parkinson's disease questionnaire in the randomized phase | up to 6 months
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the levodopa equivalent daily dose in the randomized phase | up to 6 months
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the beck depression inventory in the randomized phase | up to 6 months
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the maximal phonatory time in the randomized phase | up to 6 months
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the dysphonia severity index in the randomized phase | up to 6 months
Difference in improvement from baseline to the end of the PSA vs STN stimulation period in the Mini-Mental Status Exam in the randomized phase | up to 6 months
Adverse events | up to 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dianyou Li, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China